CLINICAL TRIAL: NCT00686049
Title: Validation of the HIV Treatment Readiness Measure (HTRM)
Brief Title: HIV Treatment-Readiness Measure (HTRM) Validation
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 065
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-02

CONDITIONS: HIV Infections
Keywords: HIV Treatment Readiness Measure (HTRM); Highly Active Antiretroviral Treatment (HAART); Adherence; Treatment readiness; HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Study Group: Participants will complete two audio computer assisted self interviews on laptop computers. This study will also involve the abstraction of participants' viral load and CD4 counts from their medical charts.

SUMMARY:
The goal of this study is to assess the reliability of the HIV

Treatment Readiness Measure (HTRM) to assist clinicians in:

(1) determining whether or not youth living with HIV are ready to initiate HAART and (2) identifying youth who may be in need of additional support services to facilitate their adherence to HAART. The current study will examine the psychometric properties of the HTRM and establish its test-retest reliability over a two week period. If the HTRM is found to be reliable, a subsequent study will examine its predictive validity.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive youth, 13 years 0 days to 24 years 364 days of age
* Either HAART naïve (defined as never having taken HAART) or HAART experienced (defined as having had at least one experience taking HAART and not having taken HAART for 30 days prior to study entry)
* Not currently on HAART, but planning to initiate HAART within the next 2 months based on provider recommendation
* Enrolled in care at an AMTU or a collaborating site
* Able to speak and understand English
* Willing to provide informed consent, or assent with parental permission (if required by the site IRB) for participation in this study.

Exclusion Criteria:

* Evidence of cognitive impairment or other mental condition that limits his/her ability to complete the assessment (per PI or designee discretion)
* Determined by the PI (or designee) to be under the influence of psychoactive agents or intoxicated at the time of assessment to a degree that would interfere with successful completion of the questionnaire
* Visibly distraught or unstable
* Any clinical condition that would likely interfere with the participant's ability to complete the study

Participants who are unable to speak English will be excluded from the initial testing of the HTRM's reliability and validity in keeping with traditional tool development strategies. If the initial study indicates that the English version of the HTRM is reliable and valid, appropriate methods will be employed to translate the instrument into Spanish and the reliability and validity will be re-examined for the Spanish version.

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: HIV-infected, English speaking youth between 13 and 24 years of age who are enrolled in care at an AMTU or collaborating site, not currently on HAART but planning to initiate HAART within the next two months.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To examine the factor structure and estimate the internal consistency of each factor of the HTRM. | 1 year
To estimate the test-retest reliability of the HTRM. | Entry, Week 2

SECONDARY OUTCOMES:
To determine an appropriate system for scoring the HTRM. | 1 year
To examine the acceptability of the HTRM. | Entry, Week 2

CONTACTS AND LOCATIONS:
Overall Officials: M. Isabel Fernández, Ph.D., Study Chair — Adolescent Trials Network
Locations (15):
- United States (14):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Childrens Diagnostic & Treatment Center, Inc, Fort Lauderdale, Florida
  - University of Miami School of Medicine, Miami, Florida
  - USF College of Medicine, Tampa, Florida
  - Ruth M Rothstein CORE Center/ John H Stroger Jr Hospital, Chicago, Illinois
  - Childrens Memorial Hospital, Chicago, Illinois
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Maryland Express Mailing Address:, Baltimore, Maryland
  - Mount Sinai Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St Jude Childrens Research Hospital, Memphis, Tennessee
- University of Puerto Rico, Medical Sciences Campus, San Juan, Puerto Rico

REFERENCES:
- See also: Adolescent Trials Network website — http://www.atnonline.org